CLINICAL TRIAL: NCT03272711
Title: Remediation of Age-related Cognitive Decline: Vortioxetine and Cognitive Training
Acronym: BBS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Queen's University (Other); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201509107
Record Dates: First submitted 2017-09-01; First posted 2017-09-05 (Actual); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Age-related Cognitive Decline
Keywords: Vortioxetine; Elderly; Online cognitive training
MeSH Terms: interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vortioxetine plus cognitive training (Experimental): Vortioxetine (10 mg) plus cognitive training 5 times weekly for 30 minutes a day
  Interventions: Drug: Vortioxetine 10 mg; Behavioral: Cognitive training program
- Placebo plus cognitive training (Placebo Comparator): Placebo plus cognitive training 5 times weekly for 30 minutes a day
  Interventions: Behavioral: Cognitive training program

INTERVENTIONS:
Drug: Vortioxetine 10 mg
  Other Names: Trintellix
  Arms: Vortioxetine plus cognitive training
Behavioral: Cognitive training program — Online training program, 30 minutes a day, 5 times a week

SUMMARY:
The purpose of this research study is to examine the potential benefits of vortioxetine in combination with at-home computerized cognitive training program to improve cognition, such as memory, attention, and concentration. This study will compare the effectiveness of vortioxetine plus cognitive training versus placebo plus cognitive training.

DETAILED DESCRIPTION:
The purpose of this research study is to examine the potential benefits of vortioxetine in combination with at-home computerized cognitive training program to improve cognition, such as memory, attention, and concentration. This study will compare the effectiveness of vortioxetine plus cognitive training versus placebo plus cognitive training.

Vortioxetine is considered investigational when used as a treatment for age-related cognitive decline, which means that it has not been approved by the U.S. Food and Drug Administration for this purpose. Vortioxetine is approved by the U.S. Food and Drug Administration as a treatment for depression, and also goes by the name Trintellix (formerly known as Brintellix). That means that, while the drug itself is approved by the FDA, it is not approved for the reasons the investigators are using it in this study.

Participation in this study entails an estimated 6 study visits over the course of approximately six months. Participants will complete various assessments at our lab at the Washington University School of Medicine along with check-in visits in-person or over the phone. Additionally, they will participate in at home computerized cognitive training for approximately six months, supplemented with either vortioxetine or placebo.

The investigators will assess memory and problem-solving abilities using paper and pencil, computerized measures, and self-assessments of how participants feel. These tests could include numbers, letters, symbols, words, or sentences. These tests will be repeated throughout the study. If eligible to do so, participants will complete a baseline MRI scan.

A subset of participants who completed a baseline MRI scan will complete another MRI scan after approximately 26 weeks of vortioxetine or placebo and at home computerized cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* Community-living men and women age 65 and older
* Age-related cognitive decline as defined by (a) self-reported cognitive dysfunction that is attributed to the aging process (in response to screening questions to the participant); (b) ability to complete cognitive battery, but still scoring less than 1 standard deviation above age-matched norms at both baseline and after the two-week cognitive training lead-in.

Exclusion Criteria:

* Known dementia or other clinical neurodegenerative illness (e.g., Parkinson's disease, cerebrovascular disease) per self-report, informant report, medical records, or neuropsychological testing
* Any current psychiatric disorder
* Medical conditions that suggest shortened lifespan, such as metastatic cancer; or would prohibit safe participation in the interventions, including cardiovascular disease or musculoskeletal conditions; or with the assessments.
* Sensory impairment that would prevent participation
* IQ < 70 as estimated by the Wechsler Test of Adult Reading
* Alcohol or substance abuse within 6 months
* Concurrent cognitive training, such as brain-training software, or other interventions expected to affect neuroplasticity
* Psychotropic medications or those with likely CNS effects (none within 4 weeks prior to study entry)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Ball K, Berch DB, Helmers KF, Jobe JB, Leveck MD, Marsiske M, Morris JN, Rebok GW, Smith DM, Tennstedt SL, Unverzagt FW, Willis SL; Advanced Cognitive Training for Independent and Vital Elderly Study Group. Effects of cognitive training interventions with older adults: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2271-81. doi: 10.1001/jama.288.18.2271. PMID 12425704
- [Background] Bowie CR, Gupta M, Holshausen K, Jokic R, Best M, Milev R. Cognitive remediation for treatment-resistant depression: effects on cognition and functioning and the role of online homework. J Nerv Ment Dis. 2013 Aug;201(8):680-5. doi: 10.1097/NMD.0b013e31829c5030. PMID 23896849
- [Background] Kozauer N, Katz R. Regulatory innovation and drug development for early-stage Alzheimer's disease. N Engl J Med. 2013 Mar 28;368(13):1169-71. doi: 10.1056/NEJMp1302513. Epub 2013 Mar 13. No abstract available. PMID 23484795
- [Background] Lampit A, Hallock H, Valenzuela M. Computerized cognitive training in cognitively healthy older adults: a systematic review and meta-analysis of effect modifiers. PLoS Med. 2014 Nov 18;11(11):e1001756. doi: 10.1371/journal.pmed.1001756. eCollection 2014 Nov. PMID 25405755
- [Derived] Lenze EJ, Stevens A, Waring JD, Pham VT, Haddad R, Shimony J, Miller JP, Bowie CR. Augmenting Computerized Cognitive Training With Vortioxetine for Age-Related Cognitive Decline: A Randomized Controlled Trial. Am J Psychiatry. 2020 Jun 1;177(6):548-555. doi: 10.1176/appi.ajp.2019.19050561. Epub 2020 Mar 26. PMID 32212856

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-nine participants were not assigned to a group. Twenty did not meet eligibility criteria for randomization, 8 individuals declined to participate further and one person was a pilot participant.
Groups:
- Vortioxetine Plus Cognitive Training: Vortioxetine (10 mg) plus cognitive training 5 times weekly for 30 minutes a day
  Vortioxetine 10 mg
  Cognitive training program: Online training program, 30 minutes a day, 5 times a week
Period: Overall Study
Arm/Group | Vortioxetine Plus Cognitive Training | Placebo Plus Cognitive Training
Started | 51 | 49
Completed | 44 | 41
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vortioxetine Plus Cognitive Training | Placebo Plus Cognitive Training | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.68 (4.77) | 71.88 (5.3) | 71.78 (5.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 23 | 26 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 50 | 48 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 40 | 38 | 78
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 51 | 49 | 100
Years of Schooling [Mean (Standard Deviation); unit: years] | 16.80 (2.48) | 16.63 (3.24) | 16.72 (2.87)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Fluid Cognitive Score
Description: Total fluid cognitive score from the NIH Toolbox as well as the speed of cognitive improvement The study utilized five cognitive tests from the NIH Toolbox Cognitive Battery that measured "fluid" cognition-the capacity for new learning and information processing. A higher score indicates indicates better performance on these tests. A total fluid cognitive score at or near 100 indicates ability that is average compared with others nationally. Scores around 115 suggest above-average fluid cognitive ability, while scores around 130 suggest superior ability. Conversely, a score around 85 suggests below-average fluid cognitive ability, and a score in the range of 70 or below suggests significant impairment.
Time Frame: Randomization (0 weeks), 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine Plus Cognitive Training | Placebo Plus Cognitive Training
Number analyzed (Participants) | 51 | 49
score on a scale
  Change in Total Fluid Cognitive Score | 6.14 (7.80) | 3.71 (7.27)
  Week 4 Total Fluid Cogntive Score | 106.06 (17.06) | 105.85 (12.38)

2. Secondary Outcome: Change in Total Fluid Cognitive Score
Description: as for outcome 1
Time Frame: Randomization (0 weeks), 4 week, 12 week, 26 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine Plus Cognitive Training | Placebo Plus Cognitive Training
Number analyzed (Participants) | 51 | 49
score on a scale
  Change at Week 4 | 6.14 (7.8) | 3.71 (7.27)
  Change at Week 12 | 8.24 (7.82) | 3.93 (6.70)
  Change at Week 26 | 7.55 (7.95) | 6.05 (8.26)
  Total Fluid Cognitive Score at Week 4 | 106.06 (17.06) | 105.85 (12.38)
  Total Fluid Cognitive Score at Week 12 | 108.12 (16.34) | 105.57 (12.31)
  Total Fluid Cognitive Score at Week 26 | 106.98 (17.19) | 107.51 (11.44)

3. Secondary Outcome: Participant Function
Description: Participant function assessed using the UCSD Performance-Based Skills Assessment (UPSA).
  A validated test that required participants to demonstrate their competence to perform everyday functioning tasks in domains such as comprehension, planning, finances, transportation and communication. A higher scores indicates a better outcome. Scores can range from a minimum of 0 to a maximum of 100.
Time Frame: Randomization (0 weeks), 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine Plus Cognitive Training | Placebo Plus Cognitive Training
Number analyzed (Participants) | 51 | 49
score on a scale
  Change in UPSA Score | 2.91 (7.26) | 1.66 (8.73)
  Total UPSA Score at Week 26 | 84.50 (8.80) | 82.44 (8.59)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Vortioxetine Plus Cognitive Training | Placebo Plus Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 2/49
Other Adverse Events (participants affected / at risk) | 31/51 | 21/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vortioxetine Plus Cognitive Training (N=51) | Placebo Plus Cognitive Training (N=49)
Worsening of Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1) — Hospitalization post bypass surgery
Hospitalization for Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine Plus Cognitive Training (N=51) | Placebo Plus Cognitive Training (N=49)
nausea (Gastrointestinal disorders) | 15 | 2
viral illness (General disorders) | 9 | 8
Rashes or pruritis (Skin and subcutaneous tissue disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 4 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 3
Dizziness (General disorders) | 3 | 0
Musculoskeletal aches (General disorders) | 3 | 3
Dental infectkons/aches (General disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03272711/Prot_SAP_000.pdf